CLINICAL TRIAL: NCT00380458
Title: Prospective, Randomized, Controlled Clinical Trial to Evaluate Recovery From Post-operative Pain in Adults After Sleep Apnea Surgery Using a Coblation Device Compared to Electrocautery
Brief Title: Study to Evaluate Recovery From Postoperative Pain After Sleep Apnea Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients enrolled. Study did not start.
Sponsor: ArthroCare Corporation (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Wendy Winters, Manager Clinical Affairs, ArthroCare Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-0406JM
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive; Sleep; Apnea; Pain; UPPP; Tonsillectomy; Narcotics
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Coblation (radiofrequency-based device)

SUMMARY:
The purpose of this study is to assess whether tonsillectomy and UPPP performed using the study device to treat Obstructive Sleep Apnea (OSA) symptoms in adults is associated with less postoperative pain during the 21-day postoperative recovery period compared to electrocautery dissection.

DETAILED DESCRIPTION:
This prospective clinical study is designed to assess whether tonsillectomy and UPPP performed using the study device to treat OSA symptoms in an adult population is associated with less postoperative pain during the 21-day postoperative recovery period compared to electrocautery dissection. The amount of post-operative pain will be assessed daily over the 21-day post-operative recovery period using two general measures: 1) self-reported pain intensity and 2) self-reported pain medication administration, including frequency of use and dose. Further, timing of self-medication will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > or = 18 years of age
* Subject has positive diagnosis of Obstructive Sleep Apnea confirmed by polysomnographic study
* Subject is a surgical candidate for UPPP and tonsillectomy with or without tongue base somnoplasty
* Subject signs IRB-approved informed consent form
* Subject is willing and able to complete required follow-up.

Exclusion Criteria:

* Subject has had a previous tonsillectomy
* Subject's RDI >40
* Subject has a history of chronic use of narcotic pain medications
* Subject is unable to take liquid opioid analgesics
* Subject requires additional surgical procedures (such as nasal septoplasty or FESS) within 28 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Number of days to cessation of narcotic pain medication use during the 21-day post-treatment period.

SECONDARY OUTCOMES:
Number of days to pain resolution as measured using a visual analogue scale during the 21-day post-treatment period.
Analysis of timing of self-administration of medication during the 21-day post-treatment period
Analysis of daily pain intensity using a visual analogue scale during the 21-day post-treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: John Bitner, MD, Principal Investigator
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Troell RJ, Powell NB, Riley RW, Li KK, Guilleminault C. Comparison of postoperative pain between laser-assisted uvulopalatoplasty, uvulopalatopharyngoplasty, and radiofrequency volumetric tissue reduction of the palate. Otolaryngol Head Neck Surg. 2000 Mar;122(3):402-9. doi: 10.1016/S0194-5998(00)70056-8. PMID 10699818
- [Background] Quinn SJ, Daly N, Ellis PD. Observation of the mechanism of snoring using sleep nasendoscopy. Clin Otolaryngol Allied Sci. 1995 Aug;20(4):360-4. doi: 10.1111/j.1365-2273.1995.tb00061.x. PMID 8548973
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Sher AE. An overview of sleep disordered breathing for the otolaryngologist. Ear Nose Throat J. 1999 Sep;78(9):694-5, 698-700, 703-6 passim. PMID 10502892